CLINICAL TRIAL: NCT01371006
Title: Effect of Multiple Dosing With 240mg q 12hrs BI 201335 on the Pharmacokinetics of 50 mg Single Dose Efavirenz and Effect of Multiple Dosing With 600mg QD Efavirenz on Cyp 3A4 and the Pharmacokinetics of BI 201335 in Healthy Volunteers
Brief Title: Evaluation of the Effect of Multiple Dosing With BI 201335 on CYP2B6 Metabolism and Effect of Multiple Dosing With Efavirenz on the Steady-state Pharmacokinetics of BI 201335 and on CYP3A4/5 Metabolism in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1220.20
Record Dates: First submitted 2011-06-09; First posted 2011-06-10 (Estimated); Results first posted 2015-08-03 (Estimated); Last update posted 2015-08-03 (Estimated); Status verified 2015-07

CONDITIONS: Healthy
MeSH Terms: interventions — Contraceptives, Oral

ARMS (2):
- BI201335 low dose Efavirenz (Experimental): low dose Efavirenz
  Interventions: Drug: low dose
- BI201335 high dose Efavirenz (Experimental): normal dose Efavirenz
  Interventions: Drug: low dose; Drug: normal dose

INTERVENTIONS:
Drug: low dose — efavirenz single dosing once daily
  Arms: BI201335 high dose Efavirenz
Drug: normal dose — efavirenz once daily
  Arms: BI201335 high dose Efavirenz
Drug: low dose — Efavirenz single dosing once daily
  Arms: BI201335 low dose Efavirenz

SUMMARY:
Obtain interaction data between BI 201335 and Efavirenz to guide dosing for each drug when administered together.

To predict drug interaction between BI 201335 and Cyp 3A4 y using Midazolam as cyp 3A4 probe , Efavirenz as enzyme inducer and BI 201335 as enzyme inhibitor.

ELIGIBILITY:
Inclusion criteria:

Healthy volunteers age 18- 55 BMI (Body Mass Index) 18.5 - 29.9

Exclusion criteria:

1. Any finding on medical examination and ECG (Electrocardiography) deviating from normal
2. Active diseases
3. History of photosensitivity or rash

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 2011-06; Primary Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- 1220.20.41001 Boehringer Ingelheim Investigational Site, Basel, Switzerland

RESULTS

PARTICIPANT FLOW:
Groups:
- Group A: 240 mg Faldaprevir+50 mg Efavirenz: Faldaprevir (soft gel capsule): Loading dose (480 mg) on day 7 followed by 240 mg doses twice a day until day 19.
  Efavirenz (film-coated tablet): Single dose (50 mg) on day 1 and 14.
  oral administration with water after food intake.
- Group B: 600 mg Efavirenz+240 mg Faldaprevir+7.5 mg Midazolam: Faldaprevir (soft gel capsule): Loading dose (480 mg) on day 2 followed by 240 mg doses twice a day until day 18.
  Efavirenz (film-coated tablet): 600 mg on days 10 to 18 once a day. Midazolam (tablet): Single dose (7.5 mg) on day 1, 9 and 18.
  oral administration with water after food intake.
Period: Overall Study
Arm/Group | Group A: 240 mg Faldaprevir+50 mg Efavirenz | Group B: 600 mg Efavirenz+240 mg Faldaprevir+7.5 mg Midazolam
Started | 14 | 15
Completed | 13 | 15
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Group B: 600 mg Efavirenz+240 mg Feldaprevir+7.5 mg Midazolam: Faldaprevir (soft gel capsule): Loading dose (480 mg) on day 2 followed by 240 mg doses twice a day until day 18.
  Efavirenz (film-coated tablet): 600 mg on days 10 to 18 once a day. Midazolam (tablet): Single dose (7.5 mg) on day 1, 9 and 18.
  oral administration with water after food intake.
- Total: Total of all reporting groups
Arm/Group | Group A: 240 mg Faldaprevir+50 mg Efavirenz | Group B: 600 mg Efavirenz+240 mg Feldaprevir+7.5 mg Midazolam | Total
Number analyzed (Participants) | 14 | 15 | 29
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.4 (10.7) | 33.1 (11.6) | 36.1 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 6 | 14
  Male | 6 | 9 | 15

OUTCOME MEASURES:

1. Primary Outcome: Group A - Efavirenz: Cmax
Description: Maximum plasma concentration (Cmax) of Efavirenz calculated for subjects in sequence group A (240 mg Faldaprevir+50 mg Efavirenz)
Time Frame: 0:00, 0:30, 1:00, 1:30, 2:00, 3:00, 4:00, 6:00, 8:00, 12:00, 24:00, 48:00, 72:00, 96:00, 120:00, 144:00 hours(h) after administration of Efavirenz
Population: all subjects entered in sequence group A of the PK set. Pharmacokinetic (PK) set: This subject set included all subjects of the treated set who provided evaluable data for at least1 observation for at least 1 primary PK endpoint in any trial period without important protocol violations.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Groups:
- 50 mg Efavirenz: single oral administration of 50 mg Efavirenz dosed alone (Day 1)
- 50 mg Efavirenz+240 mg Faldaprevir: single oral administration of 50 mg Efavirenz dosed with Faldaprevir at steady state (Day 14)
Arm/Group | 50 mg Efavirenz | 50 mg Efavirenz+240 mg Faldaprevir
Number analyzed (Participants) | 14 | 13
nmol/L | 771.0 (29.1) | 809.0 (19.9)
Statistical Analysis 1: Comparison: 50 mg Efavirenz vs 50 mg Efavirenz+240 mg Faldaprevir; relative bioavailability comparison (50 mg Efavirenz+240 mg Faldaprevir : 50 mg Efavirenz) of Efavirenz; Test type: Non-Inferiority or Equivalence — investigation of relative bioavailability (no formal testing); ANOVA; Geometric Mean Ratio = 105.61, 90% CI 2-sided [90.81 to 122.82], Standard Deviation 22.0 — the standard deviation is actually the geometric coefficient of variation

2. Primary Outcome: Group A - Efavirenz: AUC0-∞
Description: Area under the concentration-time curve of the analyte in plasma over the time interval 0 to infinity of Efavirenz calculated for subjects in sequence group A (240 mg Faldaprevir+50 mg Efavirenz)
Time Frame: 0:00, 0:30, 1:00, 1:30, 2:00, 3:00, 4:00, 6:00, 8:00, 12:00, 24:00, 48:00, 72:00, 96:00, 120:00, 144:00 h after administration of Efavirenz
Population: all subjects entered in sequence group A of the PK set.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol*h/L
Arm/Group | 50 mg Efavirenz | 50 mg Efavirenz+240 mg Faldaprevir
Number analyzed (Participants) | 14 | 13
nmol*h/L | 36100.0 (30.3) | 40700.0 (28.8)
Statistical Analysis 1: Comparison: 50 mg Efavirenz vs 50 mg Efavirenz+240 mg Faldaprevir; relative bioavailability comparison (50 mg Efavirenz+240 mg Faldaprevir : 50 mg Efavirenz) of Efavirenz; Test type: Non-Inferiority or Equivalence — investigation of relative bioavailability (no formal testing); ANOVA; Geometric Mean Ratio = 116.12, 90% CI 2-sided [101.87 to 132.35], Standard Deviation 18.8 — the standard deviation is actually the geometric coefficient of variation

3. Primary Outcome: Group B - Faldaprevir: Cmax,ss
Description: Maximum plasma concentration at steady state of Faldaprevir calculated for subjects in sequence group B (600 mg Efavirenz+240 mg Faldaprevir+7.5 mg Midazolam)
Time Frame: 0:00, 0:30, 1:00, 1:30, 2:00, 3:00, 4:00, 6:00, 8:00, 12:00 h after first administration of Faldaprevir
Population: all subjects entered in sequence group B of the PK set.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- 7.5 mg Midazolam+240 mg Faldaprevir: single oral administration of 7.5 mg Midazolam and multiple oral administration of 240 mg Faldaprevir (Day 9)
- 7.5 mg Midazolam+240 mg Faldaprevir+600 mg Efavirenz: single oral administration of 7.5 mg Midazolam and multiple oral administration of 240 mg Faldaprevir and with multiple oral administration of 600 mg Efavirenz (Day 18)
Arm/Group | 7.5 mg Midazolam+240 mg Faldaprevir | 7.5 mg Midazolam+240 mg Faldaprevir+600 mg Efavirenz
Number analyzed (Participants) | 15 | 14
ng/mL | 24000.0 (76.4) | 17200.0 (111)
Statistical Analysis 1: Comparison: 7.5 mg Midazolam+240 mg Faldaprevir vs 7.5 mg Midazolam+240 mg Faldaprevir+600 mg Efavirenz; relative bioavailability comparison (7.5 mg Midazolam+240 mg Faldaprevir+600 mg Efavirenz : 7.5 mg Midazolam+240 mg Faldaprevir) of Faldaprevir; Test type: Non-Inferiority or Equivalence — investigation of relative bioavailability (no formal testing); ANOVA; Geometric Mean Ratio = 71.83, 90% CI 2-sided [61.46 to 83.95], Standard Deviation 23.6 — the standard deviation is actually the geometric coefficient of variation

4. Primary Outcome: Group B - Faldaprevir: AUC0-12h,ss
Description: Area under the concentration-time curve of Faldaprevir at steady state over the time interval 0 to 12h calculated for subjects in sequence group B (600 mg Efavirenz+240 mg Faldaprevir+7.5 mg Midazolam)
Time Frame: 0:00, 0:30, 1:00, 1:30, 2:00, 3:00, 4:00, 6:00, 8:00, 12:00 h after first administration of Faldaprevir
Population: all subjects entered in sequence group B of the PK set.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | 7.5 mg Midazolam+240 mg Faldaprevir | 7.5 mg Midazolam+240 mg Faldaprevir+600 mg Efavirenz
Number analyzed (Participants) | 15 | 14
ng*h/mL | 225000.0 (91.1) | 146000.0 (148)
Statistical Analysis 1: Comparison: 7.5 mg Midazolam+240 mg Faldaprevir vs 7.5 mg Midazolam+240 mg Faldaprevir+600 mg Efavirenz; [analysis description as in outcome 3, analysis 1]; Test type: Non-Inferiority or Equivalence — investigation of relative bioavailability (no formal testing); ANOVA; Geometric Mean Ratio = 64.97, 90% CI 2-sided [53.32 to 79.16], Standard Deviation 30.2 — the standard deviation is actually the geometric coefficient of variation

5. Primary Outcome: Group B - Faldaprevir: C12,ss
Description: Plasma concentration 12 h after dosing of Faldaprevir at steady state calculated for subjects in sequence group B (600 mg Efavirenz+240 mg Faldaprevir+7.5 mg Midazolam)
Time Frame: 0:00, 0:30, 1:00, 1:30, 2:00, 3:00, 4:00, 6:00, 8:00, 12:00 h after first administration of Faldaprevir
Population: all subjects entered in sequence group B of the PK set.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | 7.5 mg Midazolam+240 mg Faldaprevir | 7.5 mg Midazolam+240 mg Faldaprevir+600 mg Efavirenz
Number analyzed (Participants) | 15 | 13
ng/mL | 14700.0 (119.0) | 7650.0 (277.0)
Statistical Analysis 1: Comparison: 7.5 mg Midazolam+240 mg Faldaprevir vs 7.5 mg Midazolam+240 mg Faldaprevir+600 mg Efavirenz; [analysis description as in outcome 3, analysis 1]; Test type: Non-Inferiority or Equivalence — investigation of relative bioavailability (no formal testing); ANOVA; Geometric Mean Ratio = 54.31, 90% CI 2-sided [40.47 to 72.88], Standard Deviation 44.2 — the standard deviation is actually the geometric coefficient of variation

6. Secondary Outcome: Group A - Faldaprevir: Cmax,ss
Description: Maximum plasma concentration of Faldaprevir on day 14 at steady state, calculated for subjects in sequence group A (240 mg Faldaprevir+50 mg Efavirenz)
Time Frame: 0:00, 0:30, 1:00, 1:30, 2:00, 3:00, 4:00, 6:00, 8:00, 12:00 h after administration of Faldaprevir
Population: All patients entered in sequence group A of the PK set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Group A: 240 mg Faldaprevir+50 mg Efavirenz
Number analyzed (Participants) | 13
ng/mL | 34600.0 (26.0)

7. Secondary Outcome: Group A - Faldaprevir: Tmax,ss
Description: Time of maximum concentration of Faldaprevir on day 14 at steady state, calculated for subjects in sequence group A (240 mg Faldaprevir+50 mg Efavirenz)
Time Frame: 0:00, 0:30, 1:00, 1:30, 2:00, 3:00, 4:00, 6:00, 8:00, 12:00 h after administration of Faldaprevir
Population: All patients entered in sequence sequence group A of the PK set
Measure: Median (Full Range); unit: hours
Groups:
- Group A: 240 mg Faldaprevir+50 mg Efavirenz: Faldaprevir (soft gel capsule): Loading dose (480 mg) on day 7 followed by 240 mg doses twice a day.
  Efavirenz (film-coated tablet): Single dose (50 mg) on day 1 and 14.
  oral administration with water after food intake.
Arm/Group | Group A: 240 mg Faldaprevir+50 mg Efavirenz
Number analyzed (Participants) | 13
hours | 3.00 (0.836) [2.00 to 4.03]

8. Secondary Outcome: Group A - Faldaprevir: AUC0-12h,ss
Description: Area under the concentration-time curve of Faldaprevir over the time interval 0-12h on day 14 at steady state, calculated for subjects in sequence group A (240 mg Faldaprevir+50 mg Efavirenz)
Time Frame: 0:00, 0:30, 1:00, 1:30, 2:00, 3:00, 4:00, 6:00, 8:00, 12:00 h after administration of Faldaprevir
Population: All patients entered in sequence group A of the PK set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Group A: 240 mg Faldaprevir+50 mg Efavirenz
Number analyzed (Participants) | 13
ng*h/mL | 341000 (27.2)

9. Secondary Outcome: Group A - Faldaprevir: C12,ss
Description: Plasma concentration 12 h after dosing of Faldaprevir on day 14 at steady state, calculated for subjects in sequence group A (240 mg Faldaprevir+50 mg Efavirenz)
Time Frame: 0:00, 0:30, 1:00, 1:30, 2:00, 3:00, 4:00, 6:00, 8:00, 12:00 h after administration of Faldaprevir
Population: All patients entered in sequence group A of the PK set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Group A: 240 mg Faldaprevir+50 mg Efavirenz
Number analyzed (Participants) | 13
ng/mL | 23900 (27.7)

10. Secondary Outcome: Group A - Efavirenz: Tmax
Description: Time of maximum concentration of Efavirenz on day 14, calculated for subjects in sequence group A (240 mg Faldaprevir+50 mg Efavirenz)
Time Frame: 0:00, 0:30, 1:00, 1:30, 2:00, 3:00, 4:00, 6:00, 8:00, 12:00 h after administration of Efavirenz
Population: All patients entered in sequence group A of the PK set
Measure: Median (Full Range); unit: hours
Arm/Group | Group A: 240 mg Faldaprevir+50 mg Efavirenz
Number analyzed (Participants) | 14
hours
  Day 1: Efavirenz | 3.00 (1.41) [1.50 to 4.02]
  Day 14: Efavirenz+Faldaprevir (N=13) | 3.03 [1.00 to 4.03]

11. Secondary Outcome: Group B - Faldaprevir: Tmax,ss
Description: Time of maximum concentration of Faldaprevir on Day 9 and 10 at steady state, calculated for patients in sequence group B (600 mg Efavirenz+240 mg Faldaprevir+7.5 mg Midazolam)
Time Frame: 0:00, 0:30, 1:00, 1:30, 2:00, 3:00, 4:00, 6:00, 8:00, 12:00 h after administration of Faldaprevir
Population: All patients entered in sequence group B of the PK set
Measure: Median (Full Range); unit: hours
Groups:
- Group B: 600 mg Efivirenz+240 mg Faldaprevir+7.5 mg Midazolam: Faldaprevir (soft gel capsule): Loading dose (480 mg) on day 2 followed by 240 mg doses twice a day until day 18.
  Efavirenz (film-coated tablet): 600 mg on days 10 to 18 once a day. Midazolam (tablet): Single dose (7.5 mg) on day 1, 9 and 18.
  oral administration with water after food intake.
Arm/Group | Group B: 600 mg Efivirenz+240 mg Faldaprevir+7.5 mg Midazolam
Number analyzed (Participants) | 15
hours
  Day 9: Midazolam+Faldaprevir | 3.00 [0.00 to 4.17]
  Day 18: Midazolam+Faldaprevir+Efavirenz (N=14) | 2.02 [1.00 to 4.03]

12. Secondary Outcome: Group B - Midazolam: Cmax
Description: Maximum plasma concentration of Midazolam on days 1, 9 and 18, calculated for subjects in sequence group B (600 mg Efavirenz+240 mg Faldaprevir+7.5 mg Midazolam)
Time Frame: 0:00, 0:30, 1:00, 1:30, 2:00, 3:00, 4:00, 6:00, 8:00, 12:00, 14:00, 24:00 h after administration of Midazolam
Population: all subjects entered in sequence group B of the PK set.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Groups:
- Group B: 600 mg Efivirenz+240 mg Faldaprevir+7.5 mg Midazolam: Faldaprevir (soft gel capsule): Loading dose (480 mg) on day 2 followed by 240 mg doses twice a day.
  Efavirenz (film-coated tablet): 600 mg on days 10 to 18 once a day. Midazolam (tablet): Single dose (7.5 mg) on day 1, 9 and 18.
  oral administration with water after food intake.
Arm/Group | Group B: 600 mg Efivirenz+240 mg Faldaprevir+7.5 mg Midazolam
Number analyzed (Participants) | 15
nmol/L
  Day 1: Midazolam | 110.0 (45.6)
  Day 9: Midazolam+Faldaprevir | 121.0 (46.1)
  Day 18: Midazolam+Faldaprevir+Efavirenz (N=14) | 44.9 (101.0)

13. Secondary Outcome: Group B - Midazolam: Tmax
Description: Time of maximum concentration after a single dose of Midazolam on days 1, 9 and 18, calculated for subjects in sequence group B (600 mg Efavirenz+240 mg Faldaprevir+7.5 mg Midazolam)
Time Frame: 0:00, 0:30, 1:00, 1:30, 2:00, 3:00, 4:00, 6:00, 8:00, 12:00, 14:00, 24:00 h after administration of Midazolam
Population: all subjects entered in sequence group B of the PK set.
Measure: Median (Full Range); unit: hours
Arm/Group | Group B: 600 mg Efivirenz+240 mg Faldaprevir+7.5 mg Midazolam
Number analyzed (Participants) | 15
hours
  Day 1: Midazolam | 1.00 (47.0) [0.50 to 1.50]
  Day 9: Midazolam+Faldaprevir | 1.00 (59.7) [0.50 to 3.00]
  Day 18: Midazolam+Faldaprevir+Efavirenz (N=14) | 0.74 (59.0) [0.50 to 3.02]

14. Secondary Outcome: Group B - Midazolam: AUC0-∞
Description: Area under the concentration-time curve of of Midazolam over the time interval 0 to infinity on days 1, 9 and 18, calculated for subjects in sequence group B (600 mg Efavirenz+240 mg Faldaprevir+7.5 mg Midazolam)
Time Frame: 0:00, 0:30, 1:00, 1:30, 2:00, 3:00, 4:00, 6:00, 8:00, 12:00, 14:00, 24:00 h after administration of Midazolam
Population: all subjects entered in sequence group B of the PK set.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol*h/L
Arm/Group | Group B: 600 mg Efivirenz+240 mg Faldaprevir+7.5 mg Midazolam
Number analyzed (Participants) | 15
nmol*h/L
  Day 1: Midazolam | 278 (28.3)
  Day 9: Midazolam+Faldaprevir | 624 (54.3)
  Day 18: Midazolam+Faldaprevir+Efavirenz (N=14) | 110 (88.1)

15. Secondary Outcome: Clinical Relevant Abnormalities for Vital Signs, Blood Chemistry, Haematology, Physical Examination and ECG
Description: Clinical Relevant Abnormalities for Vital Signs, Blood Chemistry, Haematology, Physical Examination and ECG. New abnormal findings or worsening of baseline conditions were reported as Adverse Events.
Time Frame: From first treatment administration (Day 1) up to Day 24
Population: treated set: All subjects who were dispensed study medication and were documented to have taken at least 1 dose of trial medication
Measure: Number; unit: participants
Arm/Group | Group A: 240 mg Faldaprevir+50 mg Efavirenz | Group B: 600 mg Efivirenz+240 mg Faldaprevir+7.5 mg Midazolam
Number analyzed (Participants) | 14 | 15
participants
  Weight decreased | 1 | 0
  Hepatic enzyme increased | 0 | 1

16. Secondary Outcome: Group A - Number of Participants With Drug Related Adverse Events
Description: Number of participants with investigator-defined drug related adverse events (AE) in sequence group A. AEs occurring up to 5 days after last intake of Faldaprevir on day 19 were assigned to Efavirenz+Faldaprevir treatment.
  AEs were assessed throughout the trial. During the outpatient portion of the trial, assessment of AEs was monitored by telephone.
Time Frame: From Day 1 up to 30 days after last treatment (Days 1,2,3,4,5,6,7,8,11,13,14,15,16,17,18,19,20,24)
Population: all subjects entered in sequence group A of the treated set.
Measure: Number; unit: participants
Groups:
- Efavirenz: Treatment with single-dose Efavirenz.
- Faldaprevir: During treatment with Faldaprevir.
- Efavirenz+Faldaprevir: During treatment with Faldaprevir and single-dose Efavirenz.
- Total On-treatment: Total number of participants with drug related adverse events during treatment.
Arm/Group | Efavirenz | Faldaprevir | Efavirenz+Faldaprevir | Total On-treatment
Number analyzed (Participants) | 14 | 14 | 13 | 14
participants | 2 | 13 | 11 | 13

17. Secondary Outcome: Group B - Number of Participants With Drug Related Adverse Events
Description: Number of participants with investigator-defined drug related adverse events (AE) in sequence group B. AEs occurring up to 5 days after last intake of Faldaprevir were assigned to Faldaprevir+Midazolam+Efavirenz treatment.
  AEs were assessed throughout the trial. During the outpatient portion of the trial, assessment of AEs was monitored by telephone.
Time Frame: From Day 1 up to 30 days after last treatment (Days 1,2,6,8,9,10,11,14,17,18,19,24)
Population: all subjects entered in sequence group B of the treated set.
Measure: Number; unit: participants
Groups:
- Midazolam: Treatment with single-dose Midazolam.
- Faldaprevir+Midazolam: During treatment with Faldaprevir and single-dose Midazolam.
- Faldaprevir+Midazolam+Efavirenz: During treatment with Faldaprevir, Efavirenz, and single-dose Midazolam
Arm/Group | Midazolam | Faldaprevir | Faldaprevir+Midazolam | Faldaprevir+Midazolam+Efavirenz | Total On-treatment
Number analyzed (Participants) | 15 | 15 | 15 | 15 | 15
participants | 1 | 14 | 3 | 14 | 15

ADVERSE EVENTS:
Time Frame: From Day 1 up to 30 days after last treatment. Group A: Days 1,2,3,4,5,6,7,8,11,13,14,15,16,17,18,19,20,24 Group B: Days 1,2,6,8,9,10,11,14,17,18,19,24
Description: AEs were assessed throughout the trial. During the outpatient portion of the trial, assessment of AEs was monitored by telephone.
Groups:
- Group A: Efavirenz: Treatment with single-dose Efavirenz in Group A.
- Group A: Faldaprevir: During treatment with Faldaprevir in Group A.
- Group A: Faldaprevir+Efavirenz: During treatment with Faldaprevir and single-dose Efavirenz in Group A.
- Group B: Midazolam: Treatment with single-dose Midazolam in Group B.
- Group B: Faldaprevir: During treatment with Faldaprevir in Group B.
- Group B: Faldaprevir+Midazolam: During treatment with Faldaprevir and single-dose Midazolam in Group B.
- Group B: Faldaprevir+Midazolam+Efavirenz: During treatment with Faldaprevir, Efavirenz, and single-dose Midazolam in Group B.
Arm/Group | Group A: Efavirenz | Group A: Faldaprevir | Group A: Faldaprevir+Efavirenz | Group B: Midazolam | Group B: Faldaprevir | Group B: Faldaprevir+Midazolam | Group B: Faldaprevir+Midazolam+Efavirenz
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/14 | 0/13 | 0/15 | 0/15 | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 3/14 | 13/14 | 11/13 | 1/15 | 14/15 | 6/15 | 15/15
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Group A: Efavirenz (N=14) | Group A: Faldaprevir (N=14) | Group A: Faldaprevir+Efavirenz (N=13) | Group B: Midazolam (N=15) | Group B: Faldaprevir (N=15) | Group B: Faldaprevir+Midazolam (N=15) | Group B: Faldaprevir+Midazolam+Efavirenz (N=15)
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rash pustular (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Abnormal dreams (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 4
Sleep disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 2
Hypnagogic hallucination (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Initial insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 3 | 0 | 0 | 4 | 0 | 10
Headache (Nervous system disorders) | 2 | 3 | 5 | 0 | 3 | 0 | 3
Circadian rhythm sleep disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Disturbance in attention (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Dysaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hyperaesthesia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ocular icterus (Eye disorders) | 0 | 4 | 0 | 0 | 5 | 1 | 0
Conjunctivitis (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 6 | 3 | 0 | 6 | 1 | 3
Diarrhoea (Gastrointestinal disorders) | 1 | 5 | 2 | 1 | 2 | 1 | 1
Vomiting (Gastrointestinal disorders) | 0 | 3 | 0 | 0 | 2 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 2 | 1 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 2
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cheilitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lip dry (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Jaundice (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 6 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 7
Rash maculo?papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Rash vesicular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Blister (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Generalised erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Renal pain (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 3
Feeling hot (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 2
Malaise (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hepatic enzyme increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Weight decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Sunburn (Injury, poisoning and procedural complications) | 0 | 0 | 4 | 0 | 1 | 0 | 0
Thermal burn (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.